CLINICAL TRIAL: NCT06517264
Title: Multicenter Clinical Trial on the Effectiveness and Safety of Outpatient Treatment of Uncomplicated Acute Diverticulitis Without Antibiotics Compared to Treatment With Antibiotics. ADIANA TRIAL
Brief Title: Effectiveness and Safety of Outpatient Treatment of Uncomplicated Acute Diverticulitis Without Antibiotics
Acronym: ADIANA
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Monica Mengual Ballester (Other)
Responsible Party: Sponsor-Investigator, Monica Mengual Ballester, Doctor in Medicine, Specialist in General and Digestive Surgery., Hospital General Universitario Morales Meseguer
Organization: Hospital General Universitario Morales Meseguer (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DIVERT-ADIANA
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Diverticulitis, Colonic
Keywords: diverticular disease; uncomplicated diverticulitis; diverticular inflammation
MeSH Terms: conditions — Diverticulitis, Colonic; Diverticular Diseases | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Intervention Model Description: Multicenter, controlled, randomized, and open-label study (without blinding) with two treatment arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Outpatient treatment with antibiotics (group A) (Active Comparator): If belonging to group A (receiving oral antibiotic therapy), the usual oral antibiotic regimen of each center will be indicated.
  According to according to the guidelines of our hospital:
  * 3rd generation cephalosporin (e.g., Cefditoren 200 mg, one tablet every 12 hours) + Metronidazole 500 mg, two tablets every 8 hours. Duration of treatment: 7 days.
  * Penicillin allergy: Ciprofloxacin 500 mg, one tablet every 12 hours + Metronidazole 500 mg, two tablets every 8 hours. Duration of treatment: 7 days.
  Hygienic-dietary measures:
  * Low-residue diet for the first 48 hours. An informative leaflet will be provided to clarify these recommendations.
  * Adequate oral hydration during the episode.
  * Paracetamol 1 gram orally, one tablet every 8 hours. If pain persists, alternate every 4 hours Paracetamol with Metamizole 575 mg, one tablet every 8 hours. If allergic to Metamizole, it can be substituted with Dexketoprofen 25 mg, one tablet every 8 hours.
  Interventions: Drug: Antibiotic
- Outpatient treatment without antibiotics (group B) (Other): Hygienic-dietary measures:
  * Low-residue diet for the first 48 hours. An informative leaflet will be provided to clarify these recommendations.
  * Adequate oral hydration during the episode.
  * Paracetamol 1 gram orally, one tablet every 8 hours. If pain persists, alternate every 4 hours Paracetamol with Metamizole 575 mg, one tablet every 8 hours. If allergic to Metamizole, it can be substituted with Dexketoprofen 25 mg, one tablet every 8 hours.
  Interventions: Other: Non antibiotic

INTERVENTIONS:
Drug: Antibiotic — antibiotic treatment, analgesics and hygienic-dietetic measures
  Other Names: Group A
  Arms: Outpatient treatment with antibiotics (group A)
Other: Non antibiotic — Analgesics and hygienic-dietetic measures
  Other Names: Group B
  Arms: Outpatient treatment without antibiotics (group B)

SUMMARY:
The objective of this clinical trial to evaluate the effectiveness and safety of outpatient treatment without antibiotics compared to outpatient treatment with antibiotics in patients with acute uncomplicated diverticulitis.

The hypotheses are:

* Null Hypothesis (H0): Outpatient treatment without antibiotics in patients with acute uncomplicated diverticulitis is neither safe nor effective and is inferior to outpatient management with antibiotics.
* Alternative Hypothesis (H1): Outpatient treatment without antibiotics in patients with acute uncomplicated diverticulitis is safe, effective, and not inferior to outpatient management with antibiotics.

We compare the rate of complications, therapeutic failure (clinical worsening and readmission) and recurrence between patients who, on an outpatient basis, are administered antibiotics and those who are not.

The patient diagnosed with acute uncomplicated diverticulitis who meets the inclusion criteria is evaluated and examined by a general surgeon. After informing him/her about the pathology, the study will be explained and he/she will be invited to freely participate in it. After accepting and signing the informed consent form, the patient will be included in the study and will be randomly assigned to one of the two treatment arms (outpatient treatment with antibiotics (group A) or without antibiotics (group B).

DETAILED DESCRIPTION:
The surgeon must reassess the patient at 72 hours, with a complete history of the new clinical status, physical examination, and blood tests (with the same parameters). This visit will check treatment adherence and early clinical response. If the patient shows unfavorable progress or clear clinical deterioration, a new imaging test will be considered, and the assigned therapeutic option will be considered a failure. Follow-up will be completed with a face-to-face consultation one month after the episode and another (face-to-face or telematic) at six months.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old with clinical and radiological diagnosis of acute sigmoid or descending colon diverticulitis (left-sided acute diverticulitis) not complicated.
* Radiological diagnosis of acute uncomplicated diverticulitis by CT (Modified Hinchey Classification 0-Ia).
* First episode or previous history of acute diverticulitis (both complicated and uncomplicated), with ≥6 months between the last episode and the current clinical presentation).
* Informed consent to participate in the study.

Exclusion Criteria:

* Age >80 years.
* Patients eligible for hospital admission and/or intravenous antibiotic therapy (at the time of diagnosis).

  * Repeated vomiting or oral intolerance.
  * Need for intravenous fluid therapy and/or close monitoring.
  * Peripheral body temperature >38ºC.
  * Deterioration of general condition and/or clinical suspicion of sepsis.
* Significant or decompensated comorbidity: ASA IV Classification (anesthetic risk of American Society of Anesthesiologists).
* Immunocompromised patients: Hematological cause, HIV with low CD4+ levels, immunosuppressive treatment, prolonged corticosteroid therapy, chemotherapy, transplanted or splenectomized patients, predisposing genetic alterations (severe combined immunodeficiency, etc.).
* Oral or intravenous antibiotic therapy 2 weeks before the onset of symptoms for another cause.
* Pregnancy.
* Inflammatory bowel disease (Crohn's disease, ulcerative colitis).
* Lack of social and home support making outpatient treatment and follow-up impossible.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effectiveness and safety of outpatient treatment without antibiotics in patients with uncomplicated diverticulitis | 1 month
  Therapeutic failure is considered when the patient reconsults before 72 hours due to unfavorable progress or clinical deterioration requiring admission.

SECONDARY OUTCOMES:
Evaluate and contrast the outcomes in terms of recurrence between outpatient treatment with and without antibiotics. | 6 months
  recurrence is defined as a new episode of diverticulitis after a period of 12 weeks without symptoms.
Evaluate and contrast the outcomes in terms of cost-effectiveness between outpatient treatment with and without antibiotics. | 6 months
  We reduce the costs derived from antibiotic treatment and its possible side effects with the same cure rates.
Study the risk factors for bad prognosis in patients with uncomplicated diverticulitis | 6 months
  Study the risk factors for diverticulitis and prognostic factors of therapeutic failure and progression to complicated diverticulitis
Evaluate the quality of life of these patients after the acute episode and the degree of satisfaction with the treatment received. | 6 months
  It will be assessed with the acute diverticulitis episode-related quality of life test (EuroQol-5D).

OTHER OUTCOMES:
Complications of diverticulitis | 6 months
  Complications are considered to be those that require admission of the patient
Mortality | 6 moths
  death caused by poor evolution of the acute process

CONTACTS AND LOCATIONS:
Locations (1):
- Monica Mengual, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bolkenstein HE, Draaisma WA, van de Wall B, Consten E, Broeders I. Treatment of acute uncomplicated diverticulitis without antibiotics: risk factors for treatment failure. Int J Colorectal Dis. 2018 Jul;33(7):863-869. doi: 10.1007/s00384-018-3055-1. Epub 2018 Apr 21. PMID 29679152
- [Result] Unlu C, de Korte N, Daniels L, Consten EC, Cuesta MA, Gerhards MF, van Geloven AA, van der Zaag ES, van der Hoeven JA, Klicks R, Cense HA, Roumen RM, Eijsbouts QA, Lange JF, Fockens P, de Borgie CA, Bemelman WA, Reitsma JB, Stockmann HB, Vrouenraets BC, Boermeester MA; Dutch Diverticular Disease 3D Collaborative Study Group. A multicenter randomized clinical trial investigating the cost-effectiveness of treatment strategies with or without antibiotics for uncomplicated acute diverticulitis (DIABOLO trial). BMC Surg. 2010 Jul 20;10:23. doi: 10.1186/1471-2482-10-23. PMID 20646266
- [Result] Hanna MH, Kaiser AM. Update on the management of sigmoid diverticulitis. World J Gastroenterol. 2021 Mar 7;27(9):760-781. doi: 10.3748/wjg.v27.i9.760. PMID 33727769
- [Result] You H, Sweeny A, Cooper ML, Von Papen M, Innes J. The management of diverticulitis: a review of the guidelines. Med J Aust. 2019 Nov;211(9):421-427. doi: 10.5694/mja2.50276. Epub 2019 Jul 28. PMID 31352692
- [Result] Francis NK, Sylla P, Abou-Khalil M, Arolfo S, Berler D, Curtis NJ, Dolejs SC, Garfinkle R, Gorter-Stam M, Hashimoto DA, Hassinger TE, Molenaar CJL, Pucher PH, Schuermans V, Arezzo A, Agresta F, Antoniou SA, Arulampalam T, Boutros M, Bouvy N, Campbell K, Francone T, Haggerty SP, Hedrick TL, Stefanidis D, Truitt MS, Kelly J, Ket H, Dunkin BJ, Pietrabissa A. EAES and SAGES 2018 consensus conference on acute diverticulitis management: evidence-based recommendations for clinical practice. Surg Endosc. 2019 Sep;33(9):2726-2741. doi: 10.1007/s00464-019-06882-z. Epub 2019 Jun 27. PMID 31250244
- [Result] Jaung R, Nisbet S, Gosselink MP, Di Re A, Keane C, Lin A, Milne T, Su'a B, Rajaratnam S, Ctercteko G, Hsee L, Rowbotham D, Hill A, Bissett I. Antibiotics Do Not Reduce Length of Hospital Stay for Uncomplicated Diverticulitis in a Pragmatic Double-Blind Randomized Trial. Clin Gastroenterol Hepatol. 2021 Mar;19(3):503-510.e1. doi: 10.1016/j.cgh.2020.03.049. Epub 2020 Mar 30. PMID 32240832
- [Result] Chabok A, Pahlman L, Hjern F, Haapaniemi S, Smedh K; AVOD Study Group. Randomized clinical trial of antibiotics in acute uncomplicated diverticulitis. Br J Surg. 2012 Apr;99(4):532-9. doi: 10.1002/bjs.8688. Epub 2012 Jan 30. PMID 22290281
- [Result] Lameris W, van Randen A, Bipat S, Bossuyt PM, Boermeester MA, Stoker J. Graded compression ultrasonography and computed tomography in acute colonic diverticulitis: meta-analysis of test accuracy. Eur Radiol. 2008 Nov;18(11):2498-511. doi: 10.1007/s00330-008-1018-6. Epub 2008 Jun 4. PMID 18523784
- [Result] van Dijk ST, Chabok A, Dijkgraaf MG, Boermeester MA, Smedh K. Observational versus antibiotic treatment for uncomplicated diverticulitis: an individual-patient data meta-analysis. Br J Surg. 2020 Jul;107(8):1062-1069. doi: 10.1002/bjs.11465. Epub 2020 Feb 19. PMID 32073652
- [Result] Mari A, Khoury T, Lubany A, Safadi M, Farraj M, Farah A, Kadah A, Sbeit W, Mahamid M. Neutrophil-to-Lymphocyte and Platelet-to-Lymphocyte Ratios Are Correlated with Complicated Diverticulitis and Hinchey Classification: A Simple Tool to Assess Disease Severity in the Emergency Department. Emerg Med Int. 2019 Aug 14;2019:6321060. doi: 10.1155/2019/6321060. eCollection 2019. PMID 31485352
- [Result] Biondo S, Golda T, Kreisler E, Espin E, Vallribera F, Oteiza F, Codina-Cazador A, Pujadas M, Flor B. Outpatient versus hospitalization management for uncomplicated diverticulitis: a prospective, multicenter randomized clinical trial (DIVER Trial). Ann Surg. 2014 Jan;259(1):38-44. doi: 10.1097/SLA.0b013e3182965a11. PMID 23732265
- [Result] Biondo S, Golda T. Enfermedad diverticular del colon. En: Parrilla P, García-Granero E, Martín E, Morales-Conde S, Navarro S, Targarona EM, editores. Cirugía AEC. 3ª edición. Madrid: Editorial Médica Panamericana, S.A; 2022. p. 547-556
- [Result] Álvarez C, Arencibia B, Balibrea del Castillo JM, Cerdán C, Dujovne P, Durán V, et al. Monografías de la AEC: Enfermedad Diverticular y Diverticulitis Aguda. Serie nº14. Madrid: Asociación Española de Cirujanos; 2022. p.15-131